CLINICAL TRIAL: NCT00536419
Title: Association Between Motorcycle Accidents, Attention Deficit/Hyperactivity Disorder and Substance Use Disorder and Motorcycle Accidents
Brief Title: Impact of Attention Deficit/Hyperactivity Disorder and Substance Use Disorder on Motorcycle Traffic Accidents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Honda do Brasil (Unknown); Novartis (Industry); Secretaria Nacional Antidrogas (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GPPG-06450
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 2 (Placebo Comparator): 4 days of placebo
  Interventions: Other: Placebo
- 1 (Experimental): MPH-SODAS at day 1 (0.3/mg/kg/day); day 2 (0.7/mg/kg/day);days 3 and 4 (1.0 mg/kg/day)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate SODAS 0.3 mg/kg/day (day 1); 0.7 mg/kg/day (day 2); 1.0 mg/kg/day (days 3 and 4)
  Arms: 1
Other: Placebo — Placebo, daily dose, 4 days, oral administration
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether motorcycle drivers with ADHD are at a greater risk for motorcycle accidents, and whether this risk can be mitigated by treatment with methylphenidate. We will evaluate the effectiveness of Methylphenidate on driving performance, among motorcycle drivers, and investigate the correlation between improvement of ADHD symptoms (inattention and impulsivity) and driving performance.

DETAILED DESCRIPTION:
Traffic accidents (car and motorcycle) are the second leading cause of death in 15-34 year-old males. Within this group, the prevalence of motorcycle accidents is currently increasing at a significantly higher rate than the prevalence of car accidents, and studies in the international literature suggest that motorcycle drivers comprise a distinct driver profile to car drivers. Motorcycles are, by design, more difficult to control, and lend themselves more to performing dangerous stunts. Mistakes and lapses in judgment are likely to have more severe consequences when motorcycles are involved, especially when one considers the exposed nature of the driver. This is of special concern in Brazil, where a large population of so called "motoboys" delivers almost everything upon request, from food to work documents.

It is well known that individuals with ADHD have more traffic problems, such as: a higher risk of a car accident; more violent crashes; more traffic violations and a greater chance of losing the driver's license. On a driving simulator, subjects with ADHD usually present with more errors and crashes, in comparison to normal controls. Treatment with Methylphenidate (MPH), however, has been shown to improve driving performance on the simulator (For example, subjects significantly reduce their speed when necessary as compared to a placebo group), and this in turn is a good indicator of better real-life driving performance.

At present, there are no studies on the effect of ADHD treatment with MPH specifically on motorcycle drivers. This is relevant, since the increasing prevalence of traffic accidents can attributed to increased incidence of motorcycle accidents. If the treatment proves effective, this study will contribute to a reduction in a major social and health concern.

ELIGIBILITY:
Inclusion Criteria:

* Professional Motorcycle Driver
* Current diagnosis of ADHD

Exclusion Criteria:

* Mental retardation
* ADHD treatment in the last month
* Psychosis

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2007-09; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Driving Performance | After 4 days of medication
ADHD symptoms (ASRS) | After 4 days of medication

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | After 4 days of medication
Adverse effects | After 4 days of medication

CONTACTS AND LOCATIONS:
Overall Officials: Luis Augusto P Rohde, MD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Claudia M Szobot, MD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Programa de Transtornos de Déficit de Atenção/Hiperatividade — http://www.ufrgs.br/prodah